CLINICAL TRIAL: NCT05112276
Title: Food4GutMarKIT - Evaluation of a Tailored Personalized Food Concept for a Healthy Gut Microbiota and Validation of Biomarkers for Monitoring of Its Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Responsible Party: Principal Investigator, Rikard Landberg, Professor, Chalmers University of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Chalmers
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Healthy, Overweight, Obese
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Diet (Active Comparator): Average Swedish diet
  Interventions: Other: Diet
- Intervention Diet (Experimental): The intervention diet will be based on food items that have shown a beneficial effect on gut microbiota associated with cardiometabolic risk factors.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — A review has been undertaken to both identify specific bacteria associated with cardiometabolic risk factors and food items that have been shown to affect such bacteria in a beneficial direction. The intervention diet will include a variety of food items e.g. vegetables, fermented vegetables, fermented dairy products and cereal products. The control diet is based on a Swedish Average Diet

SUMMARY:
The overall aim in this "proof-of-concept" study is to evaluate if a diet concept, based on foods that have individually been reported to beneficially affect gut microbiota in fact has an effect on gut microbiota composition and activity among healthy and obese subjects and whether the effects are associated with altered cardiometabolic risk factors. The aim is further to investigate if such alterations are reflected in changes of the fecal and plasma metabolome. In total, 40 men and women, who meet all the inclusion criteria and none of the exclusion criteria will be invited to participate in the study. The participants will follow an intervention diet for 6 weeks and a control diet for 6 weeks, with a 6-week wash-out period in between and will be randomized to either begin with the intervention diet or the control diet.

The study will be running over 18 weeks (including a 6-week wash-out period) and it will include 9 visits at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 18 - 70 years
* BMI 18,5-25 for normal weighed and BMI 25-39 for overweighed/obese
* Hb ≥ 120g/L
* Serum TSH <4,0 mIU/L
* Signed informed consent

Among the overweighed, they need to have waist circumference > 102 cm/88 cm for men and women respectively. All overweighed participants must have one of the following risk factors for cardiovascular decease, whereas the normal weighed could have or not elevated risk factors:

* LDL ≥ 3,0 mmol/L
* HDL ≤1.04 mmol/L
* Total cholesterol ≥ 5.0 mmol/L
* Triglycerider ≥1.69 mmol/L
* Blood pressure ≥130/85 mmHg
* Fasting glucose ≥6.1 mmol/L.

Exclusion Criteria:

* Blood donation or participation in a clinical study with blood sampling within 30 days prior to screening visit and throughout the study.
* Following any weight reduction program or having followed one during the last 6 months
* Food allergies or intolerances
* Vegetarian or other diet restrictions (due to the standardized meal plan)
* History of stomach or gastrointestinal conditions (Inflammatory bowel disease, Crohn's disease, malabsorption, colostomy, bowel resection, gastric bypass surgery etc.)
* Previous major gastrointestinal surgery
* Pregnant or lactating or wish to become pregnant during the period of the study.
* Unable to understand written and spoken Swedish
* Lack of suitability for participation in the trial, for any reason, as judged by the medical doctor or PI.
* Pharmacological medication with drugs known to affect the microbiota, e.g. antibiotics, within 6 months prior to baseline.
* Intake of probiotics within 6 months prior to baseline.
* Have type I diabetes
* Receiving pharmacological treatment for type II diabetes (treatments based on life style interventions are acceptable, as long as it is compatible with the study protocol)
* Using nicotine products on a daily basis (including chewing gum, patches, snus etc.)
* History of heart failure or heart attack (TIA) within 1 year prior to screening
* Thyroid disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Gut microbiome | 6 weeks
  Fecal samples will analyzed for composition of the gut microbiome. Difference in gut microbiota OTUs between the two diets. Baseline compared with after 6 weeks of intervention or control.
Gut microbiome | 6 weeks, 18 weeks
  Fecal samples will analyzed for composition of the gut microbiome. Change in gut microbiota OTUs between baseline and 6 and 18 weeks of intervention or control.

SECONDARY OUTCOMES:
Triglycerides | 3 weeks, 6 weeks, 12 weeks and 18 weeks
  Investigate if fasting plasma triglycerides differ between control and intervention.
Cholesterol | 3 weeks, 6 weeks, 12 weeks and 18 weeks
  Investigate if fasting plasma cholesterol differ between control and intervention.
Low-density lipid protein | 3 weeks, 6 weeks, 12 weeks and 18 weeks
  Investigate if fasting plasma Low-density lipid proteindiffer between control and intervention.
High-density lipid protein | 3 weeks, 6 weeks, 12 weeks and 18 weeks
  Investigate if fasting plasma High-density lipid protein differ between control and intervention.
Blood pressure | 3 weeks, 6 weeks, 12 weeks and 18 weeks
  Investigate if fasting blood pressure differ between control and intervention.
Fasting glucose | 3 weeks, 6 weeks, 12 weeks and 18 weeks
  Investigate if fasting plasma glucose differ between control and intervention.
C-reactive protein | 3 weeks, 6 weeks, 12 weeks and 18 weeks
  Investigate if fasting plasma C-reactive protein differ between control and intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Landberg, Dr, Principal Investigator — Chalmers University of Technology
Locations (1):
- University of Gothenburg, Department of Food and Nutrition and Sport Science, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No